CLINICAL TRIAL: NCT07316556
Title: Prospective Systematic Data Collection for Post-Marketing Surveillance of Vliwazell® Pro Wound Dressing
Brief Title: Post-Marketing Surveillance of Vliwazell® Prowound Dressing
Acronym: Vliwazell
Status: Recruiting | Type: Observational
Sponsor: Lohmann & Rauscher (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-01
Record Dates: First submitted 2025-11-28; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Acute and Chronic Wounds

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This PMCF study is conducted to confirm the effectiveness and safety of the wound dressing Vliwazell® Pro. The aim of the study is to validate the performance of Vliwazell® Pro within its intended purpose and certified indications during routine use, and to gather additional safety data. The study will examine how the use of the dressing affects the condition of the skin surrounding the wound, the wound status in terms of exudate, wound odor, and other parameters. Furthermore, the satisfaction of healthcare providers and patients with the application of the dressing will be assessed.

DETAILED DESCRIPTION:
Vliwazell® Pro is a flexible and soft superabsorbent wound dressing designed for acute and chronic wounds with moderate to very high levels of exudate (wound fluid). The inner non-woven layer helps evenly distribute the exudate and rapidly channel it into the absorbent core. Excess wound fluid is retained in this layer, protecting the wound and surrounding tissue from maceration.

Vliwazell® Pro has high absorbent capacity and reduces the need for frequent dressing changes due to saturation, allowing the wound to remain undisturbed for longer periods. The outer layer is covered with a blue non-woven fabric that shields the patient's clothing and bed linen.

ELIGIBILITY:
Inclusion Criteria:

Wound according to indication mentioned in the instructions for use:

1. Superficial acute and chronic wounds with moderate to very high amounts of exudate and that are superficial, in:

   * arterial and venous ulcers
   * diabetic ulcers
   * pressure ulcers
   * post-traumatic wounds
   * post-operative wounds healing by secondary intention
   * skin graft donor sites
   * oncological wounds
   * ulcerating tumors
   * wounds at risk of infection
   * superficial 2nd degree burns
   * lymphatic wounds
2. As secondary dressing on laparotomy wounds and fistulas or for deep wounds when used with appropriate wound filler
3. Patient has full legal capacity
4. Patient is able to understand and provide information
5. Patient has signed the written Informed Consent Form

Exclusion Criteria:

1. Age < 18 years
2. Patient with contraindication:

   * Known allergy and/or hypersensitivity to any of the product components.
   * Not for use in tunnel-forming wound pockets, as the product may expand considerably with the absorption of wound exudate.
   * Not for use on dry wounds.
3. Pregnant or lactating women
4. Patients participating in another clinical trial at the time of inclusion
5. Patient not covered by health insurance/social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators should enroll patients out of their normal patient pool. Exceptions are vulnerable patients like pregnant or lactating women, patients under 18 years or patient without full legal capacity.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Vliwazell® Pro User Satisfaction with Exudate Management | From enrollment to the end of treatment at 2 weeks
  The primary objective of this PMCF study is to assess the user satisfaction with exudate management during the use of Vliwazell® Pro.
  The primary performance parameter is defined as the proportion of users reporting a degree of satisfaction with exudate management after two weeks of treatment that is equal to or better than 4 ("acceptable"). Exudate management is assessed using a six-point Likert scale, ranging from excellent (1), very good (2), good (3), acceptable (4), poor (5), to insufficient (6). After two weeks of treatment, users will be asked to rate the exudate management using the six-level Likert scale. Treatment success is considered achieved when the mean score is equal to or better than "acceptable."

SECONDARY OUTCOMES:
Improvement of wound condition | From enrollment to the end of treatment at 2 weeks
  One secondary endpoint is the improvement of the wound condition which is measured via a six-level scale: Excellent (1), very good (2), good (3), acceptable (4), poor (5), and insufficient (6).
  During the termination visit, after two weeks of treatment with Vliwazell® Pro more than 50% of the users should rate the improvement of the wound condition as "acceptable" or better.
Safety evaluation: Incidence of maceration of wound or surrounding skin | From enrollment to the end of treatment at 2 weeks
  Monitoring of deterioration of macerated wound surrounding skin or new development of maceration. Monitoring of deterioration of macerated wound surrounding skin or new development of maceration.Maceration will be monitored via adverse event reporting. The assumption is to have less than one third (<33%; in terms of all patients) adverse events with product relationship (excluding user errors) assignable to the event maceration within the course of the study.
  Adverse events are collected via case report form AE log. AEs meeting criteria for seriousness are reported via SAE case report form and have to be reported to sponsor immediately
Safety evaluation: Incidence of skin damage due to adhesion of wound dressing | From enrollment to the end of treatment at 2 weeks.
  Monitoring of adverse events related to damage of surrounding skin caused by dressing adhesion. Allergic reactions excluded.The assumption is to have less than one third (<33%; in terms of all patients) adverse events with product relationship (excluding user errors) assignable to a damage of the skin surrounding the wound.
Safety evaluation: Incidence of bursting of wound dressing | From enrollment to the end of treatment at 2 weeks.
  Safety parameters as low bursting (adverse device effect: bursting of wound dressing) is monitored by the adverse event reporting. The assumption is that no more than 15% (in terms of all patients) adverse events with product relationship assignable to the event bursting within the course of the study.
Safety evaluation: Compatibility with other wound care products | From enrollment to the end of treatment at 2 weeks.
  Monitoring of adverse events related to use in combination with wound irrigation solutions, primary/secondary dressings, wound fillers, or retention materials.The acceptance criterion for the requirement compatibility is no more than 15% adverse events with product relationship.
Patient-reported wound pain intensity measured by NRS-11 | From enrollment to the end of treatment at 2 weeks.
  The pain felt by the patient regarding the wound and treatment of the wound is measured via the NRS-11 score. For this, the patient is asked to rate his/her level of pain on a scale from 0 (no pain) to 10 (severe pain). Two data measurements (question to the patient) are done directly before and after the treatment with Vliwazell® Pro at the visit 1/baseline visit. Last data measurements are done after the two weeks of treatment with Vliwazell® Pro at the visit 2 / termination visit
User satisfaction and usability | From enrollment to the end of treatment at 2 weeks.
  Secondary endpoint for the user satisfaction (Visit 1):
  Users will be asked at Visit 1 if the selection of sizes for the wound dressing with 10 x 10cm, 10 x 20cm, 15 x 20cm 20 x 25cm and 20 x 40cm is satisfying their needs in daily practice. This parameter is measured on a Two-Point Scale (yes/no) and the assumption (it will not be statistically tested) is that ≥50% for the answer "yes" (for each feature).
  At termination visit, users will be asked to assess predefined parameters related to dressing performance and usability. The assessment will be conducted using a six-level agreement scale:,These are measured via a six-level scale: 1- I totally agree, 2- I agree,3- Neither agree nor reject, 4- I disagree, 5-I totally disagree.
  The assumption (not statistically tested) is that as ≥50% answer: "I totally agree" or "I agree".
Patient satisfaction | From enrollment to the end of treatment at 2 weeks.
  The patient satisfaction will be collected by a quality of life (QoL) questionnaire typical for wounds. The questionnaire is asked for on initial and closed visits. On closed visit additional questions are included regarding the patient satisfaction. The patients will be asked if they think that Vliwazell® Pro is comfortable for them while wearing and whether they think that the wound dressing has a high wearing comfort. Additionally, they will be asked if clothing and bed linen are protected from soaking and if they feel protected from that by that the wound dressing.
  These parameters are measured via a six-level scale: 1- I totally agree, 2- I agree,3- Neither agree nor reject,4- I disagree, 5-I totally disagree.
  The assumption for each question is that ≥50% will answer: "I totally agree" or "I agree".

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Eberlain, Dr, Principal Investigator — Lohmann & Rauscher
Locations (8):
- Germany (8):
  - Wundmanagement, Aachen
  - MVZ Hausärzte, Brüggen
  - ORGAMed, Dortmund
  - Hautklinik, Erlangen
  - Krankenhaus Tabea, Hamburg
  - WKM Rösner Mönchengladbach, Mönchengladbach
  - Gesundheitsmanager, Inh. Christine Bertram, Waidhaus
  - WKM Rösner Willich, Willich

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy considerations and the nature of the study.